CLINICAL TRIAL: NCT04985643
Title: Local, Multicentre, Non-Interventional Study of Early Diagnostics of Multiple Myeloma Relapses Evaluation in Real Life Practice in the Russian Federation
Brief Title: A Study of Real Life Treatment for Multiple Myeloma (MM)
Acronym: LEADER
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16058
Record Dates: First submitted 2021-07-29; First posted 2021-08-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With MM: Participants diagnosed with MM (complete response [CR], very good partial response [VGPR] and partial response [PR]) and who have received one prior first line treatment within 3 months preceding the enrollment, will be observed retrospectively and medical data will be monitored and collected prospectively every 3 months until the second biochemical and symptomatic relapse is identified.

SUMMARY:
The main aim of this study is to learn how long it takes for people with MM to have a relapse after their first treatment. Not all participants will have a relapse during the study.

Participants will visit their clinic every 3 months and be treated according to their clinic's standard practice.

The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with MM relapses. This study will assess the low detection rate of biochemical relapses which will improve routine clinical practices and management of participants with MM in real world practice.

The study will enroll approximately 350 participants. The data will be collected both prospectively and/or retrospectively at the specialized care (hematology) and will be recorded into electronic case report forms (e-CRFs) of the electronic data capture (EDC) system. All the participants will be assigned to a single observational cohort:

• Participants With MM

This multi-center study will be conducted in the Russian Federation. The overall duration of the study will be approximately 4 years. The overall time for treatment and follow-up period will be approximately 2.5 years for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. With newly diagnosed multiple myeloma (NDMM) eligible and non-eligible for a high-dose therapy and autologous stem cell transplantation (HDT-ASCT) who have had a response (defined as CR, VGPR, or PR) to the ongoing SoC induction (1st line) therapy that has been started within 3 months before the inclusion.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at the time of inclusion.

Exclusion Criteria:

1. With NDMM eligible and non-eligible for a HDT-ASCT who have had SD or PD to the ongoing standard of care (SoC) induction (1st line) therapy that has been started within 3 months before the inclusion.
2. Current, previous (within the last year) or planned (for the next 15-20 months) participation in interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll participants who have a confirmed diagnosis of MM in clinical sites located in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Median Time From the Start of First Line Therapy of Participants With MM to First Biochemical Relapse of MM | From the start of the first line therapy until first biochemical relapse (up to approximately 4 years)
  According to the International Myeloma Working Group (IMWG), biochemical relapse is diagnosed in participants with relapsing MM based on the following criteria: increase in serum paraprotein by at least 25 percent (%) of nadir (absolute increase should be at least greater than or equal to [>=] 0.5 gram per liter [g/L]), increase in urine paraprotein by at least 25% (absolute increase of at least >=200 milligram per 24 hours [mg/24 h]), more than 25% increase in the difference between involved and non-involved free light chains (FLC) with abnormal FLC ratio and absolute increase of at least greater than (>) 10 milligram per deciliter (mg/dL), increase in plasmacyte infiltration by least >=10% in participants with non-secretory MM.

SECONDARY OUTCOMES:
Median Time From the Start of First Line Therapy of Participants With MM to First Biochemical Relapse of MM in the Determined Subgroups | From the start of the first line therapy until first biochemical relapse (up to approximately 4 years)
  As per IMWG, biochemical relapse diagnosed with relapsing MM on following criteria: increase in serum paraprotein by at least 25% of nadir (absolute increase should be at least >=0.5 g/L, increase in urine paraprotein by at least 25% (absolute increase of at least >=200 mg/24 h, >25% increase in difference between involved and non-involved FLC with abnormal FLC ratio and absolute increase of at least >10 mg/dL, increase in plasmacyte infiltration by least >=10% with non-secretory MM. Subgroups for analysis: MM International Staging System (ISS) stages: I, II, III; Myeloma frailty score (MFS): 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk;Best response during 1st line treatment: a PR a CR or VGPR;Performance status: Eastern Cooperative Oncology Group (ECOG) = 0-1 vs ECOG = 2;Autologous Stem Cell Transplant (ASCT) vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line
Median Time From the Start of First Line Therapy of Participants With MM | From the start of the first line therapy until first symptomatic relapse (up to approximately 4 years)
  Clinical relapse is confirmed when one or more of the following criteria (CRAB-criteria: MM-associated symptoms: hypercalcemia, renal failure, anemia, bone disease criteria). Hypercalcemia (>2.75 millimole per liter [mmol/L] or >11.5 mg/dL); renal failure: serum creatinine level >2 mg/dL (>173 mmol/L); anemia: normochromic normocytic anemia with hemoglobin level by less than (<) 2 g/dL (20 milligram per liter [mg/L]) less than the lower limit of the normal level or hemoglobin level <10 g/dL (<100 gram per liter [g/L]); bone lesions (lytic lesions, severe osteopenia, compression fractures). Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR* a CR8 or VGPR9; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers, Maintenance therapy; Treatment regimens of 1st line.
Median Time From the Start of Second Line Therapy of Participants With MM to Second Biochemical Relapse of MM | From the start of the second line therapy until second biochemical relapse (up to approximately 4 years)
  According to IMWG, biochemical relapse is diagnosed in participants with relapsing MM based on following criteria: increase in serum paraprotein by at least 25% of nadir (absolute increase should be at least >=0.5 g/L), increase in urine paraprotein by at least 25% (absolute increase of at least >=200 mg/24 h), more than 25% increase in difference between involved and non-involved FLC with abnormal FLC ratio and absolute increase of at least >10 mg/dL, increase in plasmacyte infiltration by least >=10% in participants with non-secretory MM. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line;Therapeutic regimens of 2nd line (Rd, VRD, KRd, IxaRd, DaraRd, EloRd, other).
Median Time From the Start of Second Line Therapy of Participants With MM to Second Symptomatic Relapse of MM | From the start of the second line therapy until second symptomatic relapse (up to approximately 4 years)
  Clinical relapse is confirmed when one or more of the following criteria (CRAB-criteria: MM-associated symptoms, including hypercalcemia, renal failure, anemia, bone disease criteria) are found. Hypercalcemia (>2.75 mmol/L or >11.5 mg/dL), renal failure: serum creatinine level >2 mg/dL (>173 mmol/L), anemia: normochromic normocytic anemia with hemoglobin level by <2 g/dL (20 mg/L) less than the lower limit of the normal level or hemoglobin level <10 g/dL (<100 g/L), bone lesions (lytic lesions, severe osteopenia, compression fractures). Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line;Therapeutic regimens of 2nd line (Rd, VRD, KRd, IxaRd, DaraRd, EloRd, other).
PFS1L: Progression-free Survival (PFS) From the Start of first Line Therapy to the First Biochemical Relapse | From the start of the first line therapy until first significant biochemical relapse or until the disease progression or death due to any reason whichever occurs first (up to approximately 4 years)
  PFS1L:interval from start of 1st line therapy to 1st significant biochemical relapse. As per IMWG, biochemical relapse diagnosed in participants with relapsing MM on following criteria: increase in serum paraprotein by at least 25% of nadir (absolute increase should be at least >=0.5 g/L, increase in urine paraprotein by at least 25% (absolute increase of at least >=200 mg/24 h, >25% increase in difference between involved and non-involved FLC with abnormal FLC ratio and absolute increase of at least >10 mg/dL, increase in plasmacyte infiltration by least >=10% with non-secretory MM. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
PFS2L: Progression-free Survival From the Start of Second Line Therapy to the Second Biochemical Relapse | From the start of the second line therapy until second significant biochemical relapse or until the disease progression or death due to any reason whichever occurs first (up to approximately 4 years)
  PFS2L: interval from start of 2nd line therapy to 2nd significant biochemical relapse. As per IMWG, biochemical relapse diagnosed in participants with relapsing MM on following criteria: increase in serum paraprotein by at least 25% of nadir (absolute increase should be at least >=0.5 g/L, increase in urine paraprotein by at least 25% (absolute increase of at least >=200 mg/24 h, >25% increase in difference between involved and non-involved FLC with abnormal FLC ratio and absolute increase of at least >10 mg/dL, increase in plasmacyte infiltration by least >=10% with non-secretory MM. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line;Therapeutic regimens of 2nd line (Rd, VRD, KRd, IxaRd, DaraRd, EloRd, other).
DOT1: Duration of the First Line Therapy | From initiation of the first drug to discontinuation of the last drug in the frame of first line therapy (approximately 4 years)
  DOT1 is defined as time from initiation of the first drug to discontinuation of the last drug in the frame of first line of therapy. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
DOMT1: Duration of 1st Line Maintenance Therapy | From initiation of the first line maintenance therapy to discontinuation of the last drug in the frame of first line maintenance therapy (approximately 4 years)
  DOMT1 is defined as the treatment duration of first line maintenance therapy. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
DOT2: Duration of the Second Line Therapy | From initiation of the first drug to discontinuation of the last drug in the frame of second line therapy (approximately 4 years)
  DOT2 is defined as time from initiation of the first drug to discontinuation of the last drug in the frame of second line of therapy. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line;Therapeutic regimens of 2nd line (Rd, VRD, KRd, IxaRd, DaraRd, EloRd, other).
PR1L: Percentage of Participants With Partial Response After First Line Therapy | From the end of the first line therapy up to approximately 4 years
  PR is defined as >=50% reduction of serum M protein and >=90% or <200 mg reduction urinary M protein in 24-hour, or >50% decrease in difference between involved and uninvolved FLC levels, or >50% reduction in bone marrow plasma cells, if bone marrow plasma cells >30% and >50% reduction in size of soft tissue plasmacytomas at baseline. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
VGPR1L: Percentage of Participants With VGPR After First Line Therapy | From the end of the first line therapy up to approximately 4 years
  VGPR defined as >90% reduction (<100 mg/24-hour) in serum M-protein + urine M-protein detectable by immunofixation but not on electrophoresis. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
CR1L: Percentage of Participants With Complete Response After First Line Therapy | From the end of the first line therapy up to approximately 4 years
  Complete response is defined as >5% plasma cells in myelogram with absence of paraprotein in serum and urine according to immunofixation. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line.
ORR2L: Percentage of Participants With Objective Response Rate After the Second Line Therapy | From the end of the second line therapy up to approximately 4 years
  ORR2L: percentage of participants with CR, VGPR or PR assessed by IMWG to 2nd line therapy. Per IMWG criteria, CR: >5% plasma cells in myelogram with absence of paraprotein in serum and urine according to immunofixation; VGPR: >90% reduction (<100 mg/24-h) in serum M-protein + urine M-protein detectable by immunofixation but not on electrophoresis; PR: >=50% reduction of serum M protein and >=90% or <200 mg reduction urinary M protein in 24-hour, or >50% decrease in difference between involved and uninvolved FLC levels, or >50% reduction in bone marrow plasma cells, if bone marrow plasma cells >30% and >50% reduction in size of soft tissue plasmacytomas at baseline. Subgroups for analysis: MM ISS stages: I, II, Ill; MFS: 0 and 1 vs 2 and more;Cytogenetic high-risk vs standard risk; Best response during 1st line treatment;ECOG = 0-1 vs 2, ASCT vs non-ASCT receivers;Maintenance therapy;1st and 2nd line Treatment regimens.
SD2L: Percentage of Participants With Stable Disease After the Second Line Therapy | From the end of second line therapy up to approximately 4 years
  Stable disease (SD) is defined as any state that does not meet PR, VGPR, CR, or progressive disease (PD) criteria. Subgroups for analysis: MM ISS stages: I, II, III; MFS: 0 and 1 vs 2 and more;Cytogenetic risk: high-risk vs standard risk; Best response during 1st line treatment: a PR a CR or VGPR; Performance status: ECOG = 0-1 vs ECOG = 2, ASCT vs non-ASCT receivers; Maintenance therapy; Treatment regimens of 1st line;Therapeutic regimens of 2nd line (Rd, VRD, KRd, IxaRd, DaraRd, EloRd, other).
PD2L: Percentage of Participants With Progressive Disease After Second Line Therapy | From the end of second line therapy up to approximately 4 years
  PD: increase in M-gradient by >=25% of least achieved serum (increase by >=5 g/L), urine (increase by >=200 mg/24 h) levels. With disease, "unmeasurable" by standard immunochemistry, but "measurable" by FLC level, progression: stated with increase in difference between involved and non-involved FLC by 100 mg/L. Progression: increase in bone marrow plasmatic cells level (absolute count-not less than by 10%), occurrence of new bone lesions or increase in size of previously detected ones, occurrence of new soft tissue plasmocytomas or increase in its size, hypercalcemia (corrected serum calcium level >11.5 mg/dL or 2.65 mmol/L) may be related to proliferation. Subgroups for analysis: MM ISS stages: I, II, Ill; MFS: 0 and 1 vs 2 and more;Cytogenetic high-risk vs standard risk; Best response during 1st line treatment;ECOG = 0-1 vs 2, ASCT vs non-ASCT receivers;Maintenance therapy;1st and 2nd line Treatment regimens.
Percentage of Participants With High-risk Cytogenetic Disorders at the Time of the First Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (up to approximately 4 years)
  High-risk Cytogenetic Disorder is defined as risk according to cytogenetic profile at relapse (t[4;14], del (17p), amp (1q21), hypodiploidy) at the time of the first symptomatic relapse.
Percentage of Participants With High β2-microglobulin (ß2M) or Low Albumin Levels at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
  ß2M levels is defined as >5.5 mg/L and low albumin levels is defined as <3.5 g/dL at first symptomatic relapse.
Percentage of Participants With Extramedullary Lesions at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
Percentage of Participants With Lactate Dehydrogenase (LDH) Levels Above Normal at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
Percentage of Participants With Short Duration of Response or PD During Therapy at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
  PD is defined as increase in M-gradient by >=25% of least achieved serum (increase by >=5 g/L), urine (increase by >=200 mg/24 h) levels. For participants with disease, "unmeasurable" by standard immunochemistry, but "measurable" by FLC level, progression is stated with increase in difference between involved and non-involved FLC by 100 mg/L. Progression is also indicated by increase in bone marrow plasmatic cells level (absolute count - not less than by 10%), occurrence of new bone lesions or increase in size of previously detected ones, occurrence of new soft tissue plasmocytomas or increase in it's size, hypercalcemia (corrected serum calcium level >11.5 mg/dL or 2.65 mmol/L) that may be related to proliferation. Short duration of response <6 months.
Percentage of Participants With Circulating Plasma Cells at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
Percentage of Participants With ISS stages II/III at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
  ISS is a measuring scale having three stages Stage I:low risk, β2-Microglobulin <3.5mg/L and albumin >=3.5g/dL, Stage II: not stage I or III, Stage III: high risk,β2-Microglobulin >=5.5mg/L.
Percentage of Participants With Isotypic Transformation at the Time of the First and Second Symptomatic Relapse | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
  Isotypic Transformation is defined as change in the type of secretion of light chains, hypersecretory disease.
Percentage of Participants With First and Second Symptomatic Relapse who Have Aggressive Clinical Disease Manifestations | From the start of the first line therapy until first symptomatic relapse (for first symptomatic relapse) and until second symptomatic relapse (for second symptomatic relapse) (up to approximately 4 years)
  Aggressive clinical disease manifestations include the rapid development/quick start of symptoms manifestations, an advanced diseases stages based on the laboratory results, radiography or pathomorphological examinations, organ failure (disease-related organ disorder).
Number of Participants Reporting One or More Adverse Events (AEs) With First Line Therapy | Up to approximately 4 years
Number of Participants Reporting One or More AEs With Second Line Therapy | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (24):
- Russia (24):
  - Altai Regional Clinical Hospital, Barnaul, Altayskiy Kray
  - Kaluga Regional Clinical Hospital, Kaluga, Central Federal District
  - Smolensk Clinical Hospital of Russian Railways-Medicine, Smolensk, Central Federal District
  - City Clinical Hospital No. 1 named after prof. S.I.Sergeev, Khabarovsk, Far Eastern Federal District
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov, Kirov Oblast
  - GUZ "Lipetsk City Hospital No. 3" Free Falcon ", Lipetsk, Lipetsk Oblast
  - National Research Center of Hematology of the Ministry of Health, Moscow, Moscow Oblast
  - Herzen Moscow Scientific Research Oncological Institute, Moscow, Moscow Oblast
  - Moscow Regional Research Clinical Institute n.a. M.F. Vladimirsky, Moscow, Moscow Oblast
  - BaltikMed Clinic, Kaliningrad, Northwestern Federal District
  - Vologda Regional Clinical Hospital, Vologda, Northwestern Federal District
  - Novosibirsk State Medical University, Department of Therapy, Hematology and Transfusiology based on City Clinical Hospital No. 2, Novosibirsk, Novosibirsk Oblast
  - Orenburgskaya Regional Clinical Hospital n.a. V.I. Voinova, Orenburg, Orenburgskaya District
  - Republican hospital named after V.A.Baranov, Petrozavodsk, Republic of Karelia
  - Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan, Kazan', Republic Tatarstan
  - City Clinical Hospital No. 31, Saint Petersburg, Sankt-Peterburg
  - Razumovskiy Saratov State Medical University, University Clinical, Saratov, Saratov Oblast
  - Tomsk Regional Clinical Hospital, Tomsk, Siberian Federal District
  - District Clinical Hospital, Khanty-Mansiysk, Tyumen Oblast
  - Surgut Regional Clinical Hospital, Surgut, Tyumen Oblast
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - City Clinical Hospital No. 12, Nizhny Novgorod, Volga Federal District
  - Clinic Akademicheskaya LLC, Volgograd, Volgogradskaya District
  - Republican Clinical Hospital named after G.G. Kuvatov, Ufa

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/611151a5cd353f0032b92051